CLINICAL TRIAL: NCT03080688
Title: Prizma Pulse Oximeter Evaluation
Status: Completed | Type: Observational
Sponsor: G Medical Innovations Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BYL20160415
Record Dates: First submitted 2017-02-27; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Prizma: Measurement of oxyhemoglobin saturation by OSM-3 oximeter and Prizma oxygen saturation measurement
  Interventions: Device: Prizma Oxygen Saturation Measurement

INTERVENTIONS:
Device: Prizma Oxygen Saturation Measurement — A radial arterial cannula was placed in either the left or right wrist of each subject.
  Blood gas analysis to determine oxyhemoglobin saturation was performed on an OSM-3® multi-wavelength oximeter (Hemoximeter, Radiometer, Copenhagen). No subject was anemic (Hemoglobin ≤ 10gm•dl-1).

SUMMARY:
This study is intended to evaluate performance of the new design sufficiently to support performance claims for an FDA 510K submission or ISO technical file. Specifically:

* SpO2 value range 70% to 100%
* 10 or more subjects, at least 3 of dark pigmentation
* At least 200 data points
* Meeting the following test required by the 2013 FDA Guidance on Pulse Oximeters - Premarket Notification Submissions and by ISO 80601-2-61 on Pulse Oximeters:
* 2013 FDA Guidance on Pulse Oximeters - Premarket Notification Submissions:

  * 4.1. ACCURACY OF PULSE OXIMETERS
  * 4.1.1 IN VIVO TESTING FOR SPO2 ACCURACY UNDER LABORATORY CONDITIONS
* ISO 80601-2-61:2011 Annex EE.2 and clause 201.12.1.101.2

  * 201.12.1.101 SpO2 accuracy of pulse oximeter equipment
  * 201.12.1.101.2 Determination of SpO2 accuracy

DETAILED DESCRIPTION:
The device under test was the Prizma which is a phone cover biometric device that includes reflectance oximetry. This device is a spot checker that requires the patient to hold their finger on the sensor during the measurement. The subjects were asked not to move during the study. In order to get consistent measurements the fingers were taped to the test device. The tape acted mainly as a reminder, and there were some problems with finger movement. A radial arterial cannula was placed in either the left or right wrist of each subject.

Blood gas analysis to determine oxyhemoglobin saturation was performed on an OSM-3® multi-wavelength oximeter (Hemoximeter, Radiometer, Copenhagen). No subject was anemic (Hemoglobin ≤ 10gm•dl-1). Each subject had control data taken at the beginning of each experiment, with two control blood samples drawn while breathing room air. Hypoxia was induced to different levels of oxyhemoglobin saturation (between 70-100%) by having subjects breathe mixtures of nitrogen, room air, and carbon dioxide. Oxyhemoglobin saturation was reduced to a series of targets and stabilized at the plateau value. Each plateau level of oxyhemoglobin saturation was maintained for at least 30 seconds. Two arterial blood samples were then obtained, approximately 30 seconds apart. A total of 24 samples were obtained per subject. Data were recorded by Bickler-Ye lab and provided for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects
* Healthy subjects capable of undergoing controlled hypoxemia to the levels outlined in the desaturation profile below.
* Meeting the demographic requirements listed above.

Exclusion Criteria:

* Smokers or individuals exposed to high levels of carbon monoxide that result in carboxyhemoglobin levels over 3% as tested by the BYL.
* Subjects who would be placed under medical risk under the desaturation profile listed below.
* Significant arrhythmia
* Age below 21 or over 50
* Pregnant women

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Selection of patients, both male and female, who meet the eligibility criteria (see below)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-16 (Actual)

PRIMARY OUTCOMES:
Blood oxygen saturation | 2 days
  Comparison of Measurements: Prizma Device versus Gold Standard

IPD SHARING:
Plan to Share IPD: No